CLINICAL TRIAL: NCT01782482
Title: A Comparison of Two Color Contact Lenses in Habitual Clear Contact Lens Wearers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: C-12-003
Record Dates: First submitted 2013-01-31; First posted 2013-02-04 (Estimated); Results first posted 2014-03-28 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-03

CONDITIONS: Myopia; Refractive Error
Keywords: Color contact lenses; Refractive error; Myopia
MeSH Terms: conditions — Myopia; Refractive Errors

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- AIR OPTIX® COLORS (Experimental): Lotrafilcon B contact lens with color worn on a daily wear basis for 7 days. Lenses were worn bilaterally for a minimum of 5 days per week, 8 hours per day.
  Interventions: Device: Lotrafilcon B contact lens with color
- FRESHLOOK® COLORBLENDS (Active Comparator): Phemfilcon A contact lens with color worn on a daily wear basis for 7 days. Lenses were worn bilaterally for a minimum of 5 days per week, 8 hours per day.
  Interventions: Device: Phemfilcon A contact lens with color

INTERVENTIONS:
Device: Lotrafilcon B contact lens with color — Silicone hydrogel contact lens with color
  Other Names: AIR OPTIX® COLORS
  Arms: AIR OPTIX® COLORS
Device: Phemfilcon A contact lens with color — Hydrogel contact lens with color
  Other Names: FRESHLOOK® COLORBLENDS
  Arms: FRESHLOOK® COLORBLENDS

SUMMARY:
The purpose of this study was to evaluate overall satisfaction with AIR OPTIX® COLORS as compared to FRESHLOOK® COLORBLENDS contact lenses.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to sign Informed Consent Document. If under legal age of consent, legally authorized representative must also sign Informed Consent Document.
* Able to achieve best corrected visual acuity (BCVA) of 20/25 (Snellen) or better in each eye at distance.
* Manifest cylinder less than or equal to 0.75 diopter in each eye.
* Wear contact lenses within protocol-defined specifications.
* Require spherical contact lenses within the available range of powers.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Any eye condition that contraindicates contact lens wear.
* Any systemic or ocular abnormality, infection, or disease likely to affect successful wear of contact lenses or use of their accessory solutions.
* Moderate or severe ocular findings upon examination.
* Any use of systemic or ocular medications that could contraindicate contact lens wear, including use of topical ocular medications requiring instillation during contact lens wear, except for approved lubricating drops.
* Habitual lenses worn in an extended wear modality (routinely sleeping in lenses overnight for 1 night per week or more) over the last 3 months prior to enrollment.
* Previous corneal or refractive surgery or irregular cornea.
* Eye injury or surgery within the last 6 months (excluding placement of punctal plugs).
* Monovision and monocular subjects (only one eye with functional vision) or subjects fit with only one lens.
* History of intolerance or hypersensitivity to any component of the test articles.
* Other protocol-defined exclusion criteria may apply.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 574 (Actual)
Dates: Start 2013-02; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Holden Thomas, O.D., Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 30 study centers, located in the United States.
Pre-assignment Details: Of the 574 enrolled, 13 participants did not meet all inclusion/exclusion criteria and were exited as screen failures. This reporting group includes all enrolled and randomized participants (561).
Period: Overall Study
Arm/Group | AIR OPTIX® COLORS | FRESHLOOK® COLORBLENDS
Started | 281 | 280
Completed | 271 | 270
Not Completed | 10 | 10
Not completed — Adverse Event | 2 | 1
Not completed — Lost to Follow-up | 2 | 3
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Randomized in Error | 2 | 2
Not completed — Habitually wearing toric lens OS | 0 | 1

BASELINE CHARACTERISTICS:
Population: The analysis population includes all randomized participants who satisfied specific Inclusion/Exclusion Criteria, did not sleep overnight in study lenses, and used only the habitual lens care during the study (552).
Groups:
- Total: Total of all reporting groups
Arm/Group | AIR OPTIX® COLORS | FRESHLOOK® COLORBLENDS | Total
Number analyzed (Participants) | 278 | 274 | 552
Age, Customized [Number; unit: participants]
  16-17 years | 11 | 11 | 22
  18-64 years | 267 | 263 | 530
  ≥65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 247 | 254 | 501
  Male | 31 | 20 | 51

OUTCOME MEASURES:

1. Primary Outcome: Subjective Rating of Overall Satisfaction
Description: Overall satisfaction, as rated by the participant on a 10-point scale, with 1 being very dissatisfied to 10 being very satisfied. The participant rated both eyes together by providing one single rating.
Time Frame: Day 7
Population: The analysis population includes all randomized participants who satisfied specific Inclusion/Exclusion Criteria, did not sleep overnight in study lenses, and used only the habitual lens care during the study. The actual sample size used in calculating the outcome measure may be smaller due to missing responses and/or visit attendance.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | AIR OPTIX® COLORS | FRESHLOOK® COLORBLENDS
Number analyzed (Participants) | 278 | 274
Units on a scale | 7.45 (0.17) | 6.91 (0.17)

2. Secondary Outcome: Positive Purchase Intent
Description: As reported on a questionnaire in response to, "Assuming these lenses were at a price you would expect to pay, how likely would you be to purchase these lenses?" The binary 'positive' vs 'negative' response variable was derived from a 5-point Likert scale. Positive purchase intent is reported as the percentage of participants choosing "Definitely would purchase" or "Probably would purchase."
Time Frame: Day 7
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | AIR OPTIX® COLORS | FRESHLOOK® COLORBLENDS
Number analyzed (Participants) | 278 | 274
Percentage of participants | 51.7 | 42.5

ADVERSE EVENTS:
Time Frame: Adverse Events (AE) were collected for the duration of the study (2 months). AEs were obtained as solicited comments and as observations by the study Investigator.
Description: The analysis population includes all participants/eyes exposed to the study products. 5 participants from Test (AIR OPTIX® COLORS) and 6 participants from Control (FRESHLOOK® COLORBLENDS) were randomized but not exposed to the investigational products. Color selection and/or trial-fitting lenses were not considered study products.
Arm/Group | AIR OPTIX® COLORS | FRESHLOOK® COLORBLENDS
Serious Adverse Events (participants affected / at risk) | 0/276 | 0/274
Other Adverse Events (participants affected / at risk) | 0/276 | 0/274

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.